CLINICAL TRIAL: NCT06293664
Title: Randomized Cross-over Designed Study of the Physiological Impact of Alpha MSH on Glycemic Response to an Oral Glucose Tolerance Test in Patients With Type 2 Diabetes
Brief Title: Protocol for Alpha MSH Infusion Study in Patients With Type 2 Diabetes
Acronym: α-MSH & T2DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, CMO, Dasman Diabetes Institute
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Screening
Other Study IDs: RAHM-2023-006
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes, Alpha-melanocyte stimulatory hormone (ɑ-MSH), OGTT
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The research involves a double-blinded, randomized, placebo-controlled crossover study to assess the therapeutic potential of α-MSH infusion in T2DM patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- α-MSH infusion (Experimental): Pharmaceutical grade α-MSH will be dissolved in 0.9% saline containing 0.5% human albumin.
  Interventions: Other: α-MSH infusion
- Saline infusion (Placebo Comparator): Saline infusion: Pharmaceutical GMP-grade sterile 0.5% human albumin dissolved in saline.
  Interventions: Other: Placebo solutions

INTERVENTIONS:
Other: α-MSH infusion — Pharmaceutical grade α-MSH is custom synthesized to GMP standards by Auspep (Australia www.auspep.com.au), a good manufacturing practice (GMP) accredited manufacturer of peptides, approved by the Therapeutic Goods Administration (TGA), European Medicines Agency (EMA) and U.S. Food and Drug Administration (FDA).
  Arms: α-MSH infusion
Other: Placebo solutions — Pharmaceutical GMP-grade sterile 0.5% human albumin dissolved in saline.
  Arms: Saline infusion

SUMMARY:
Alpha-melanocyte stimulatory hormone (α-MSH) is a melanocyte-stimulating hormone produced by the hypothalamus and released from the pituitary gland. It acts as an agonist to the melanocortin 5 receptor (MC5R) in human skeletal muscle, playing a role in glucose uptake and disposal. This study aims to investigate whether α-MSH can enhance glucose tolerance in patients with Type 2 Diabetes Mellitus (T2DM).

DETAILED DESCRIPTION:
Pre-clinical studies in mice have shown improved glucose clearance with α-MSH infusion, particularly in skeletal muscle. Research has demonstrated that α-MSH improves glucose tolerance in healthy humans by promoting glucose uptake in skeletal muscle cells.

Therefore this study seeks to answer the question of whether alpha-MSH improves glucose tolerance in patients with T2DM. This will be addressed through measuring the impact of α-MSH infusion in patients with T2DM. The research involves a double-blinded, randomized, placebo-controlled crossover study.

ELIGIBILITY:
Inclusion Criteria:

* People with T2DM treated with oral or injectable medications which have been stable for 3 months, but not insulin therapy for type 2 diabetes.
* Stable body weight and HbA1c for at least 3 months
* The participant is capable of giving written informed consent
* The participant is able to read, comprehend and record information written in English

Exclusion Criteria:

* Previous or current psychiatric diagnosis listed in DSM-V Axis 1.
* Significant current or past medical or psychiatric history that, in the opinion of the investigators, contraindicates their participation.
* History of type 1 diabetes mellitus.
* History of endocrine disorder.
* History of ischaemic heart disease, hypertension (current BP > 160/95 mmHg), heart failure, cardiac arrhythmia, peripheral vascular or cerebrovascular disease.
* History or presence of significant respiratory, gastrointestinal, hepatic, oncological, neurological or renal disease or other condition that in the opinion of the Investigators may affect participant safety or outcome measures.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History of sensitivity to any of the peptides, or components thereof, or a history of drug or other allergy that, in the opinion of the investigators, contraindicates their participation.
* Use of current regular prescription or over-the-counter medications that in the opinion of the Investigators may affect participant safety or outcome measures.
* Clinically significant abnormalities in screening electrocardiogram (ECG) or blood tests abnormalities which in the opinion of the study physician, is clinically significant and represents a safety risk.
* Current pregnancy or breast-feeding in female participants (the investigators would advise using contraception for the duration of the study).
* Pulse rate <40 or >100 beats per minute OR systolic blood pressure >160 and <100 and a diastolic blood pressure >95 and <50 in the semi-supine position.
* The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first experimental visit in the current study: 90 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than 3 new investigational medicinal products within 12 months prior to the screening.
* Participants who have donated, or intend to donate, blood within three months before the screening visit or following study visit completion.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2024-04-04 (Estimated); Study Completion 2024-04-04 (Estimated)

PRIMARY OUTCOMES:
Difference in the total or incremental area under the curve of glucose and insulin concentration at an OGTT during saline vs. α-MSH infusion | 12 months

SECONDARY OUTCOMES:
Difference in the total or incremental area under the curve of the concentration of metabolites (C-peptide, Glucagon, Gut hormones, α-MSH) during OGTT with saline or α-MSH infusion. | 12 months

OTHER OUTCOMES:
Difference in energy intake measured by an ad libitum meal test at the saline vs. α-MSH infusion | 12 months
Adverse events (including flushing) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided